CLINICAL TRIAL: NCT05070390
Title: An Open-Label Clinical Study to Evaluate the Pharmacokinetics of MK-0616 Following Administration of a Single Dose to Participants With Moderate Renal Impairment
Brief Title: A Study of Enlicitide Chloride (MK-0616 Oral PCSK9 Inhibitor) in Participants With Moderate Renal Impairment (MK-0616-007)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 0616-007; MK-0616-007 (Other: Merck)
Record Dates: First submitted 2021-10-01; First posted 2021-10-07 (Actual); Results first posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Moderate Renal Impairment
MeSH Terms: interventions — MK-0616

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Panel A - Moderate Renal Impairment (RI) (Experimental): Single dose of enlicitide chloride 10 mg
  Interventions: Drug: Enlicitide Chloride
- Panel B - Healthy Controls (Experimental): Single dose of enlicitide chloride 10 mg
  Interventions: Drug: Enlicitide Chloride

INTERVENTIONS:
Drug: Enlicitide Chloride — 10 mg capsule administered orally
  Other Names: MK-0616

SUMMARY:
This study evaluated the safety, tolerability and pharmacokinetic (PK) effects of enlicitide chloride in participants with moderate renal impairment (RI) to those of healthy matched control participants. Moderate RI was defined as the estimated glomerular filtration rate (eGFR) ≥30 and <60milliliter/minute/1.73meters^2 (ml/min/1.73m^2). There is no formal hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Good health based upon medical history, physical examination, vital signs, laboratory safety tests, and electrocardiograms (ECG) performed before randomization
* Body mass index (BMI) ≥18 kg/m^2 and ≤40 kg/m^2
* Male participants must agree to the following during the intervention period and for at least 90 days after the last dose of study intervention: Refrain from donating sperm, PLUS either be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent, or use acceptable contraception per study protocol
* Female participants must be of non-childbearing potential
* Moderate RI participants: Baseline estimated glomerular filtration rate (eGFR) ≥30 and <60 mL/min/1.73 m^2 based on the Modification of Diet in Renal Disease (MDRD) equation
* Moderate Renal Impairment (RI) participants: No clinically significant change in renal status at least 1 month prior to dosing and not currently receiving or has not previously been on hemodialysis
* Healthy Matched Controls: eGFR ≥80 mL/min/1.73 m^2 based on the MDRD equation

Exclusion Criteria:

* Healthy Matched Controls: history of clinically significant endocrine, GI, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Mentally or legally incapacitated, has significant emotional problems at the time of prestudy (screening) visit or expected during the conduct of the study or has a history of clinically significant psychiatric disorder of the last 5 years. Participants who have had situational depression may be enrolled in the study at the discretion of the investigator
* History of cancer, with the exception of adequately treated nonmelanomatous skin carcinoma or carcinoma in situ of the cervix or other malignancies that have been successfully treated with appropriate follow up and therefore unlikely to recur for the duration of the study
* History of significant multiple and/or severe allergies
* Positive for hepatitis B surface antigen (HBsAg), hepatitis C antibodies or human immunodeficiency virus (HIV)
* History of major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the prestudy (screening) visit
* Moderate RI participants: Does not agree to follow the smoking restrictions as defined by the study
* Healthy Matched Controls: History of smoking and/or has used nicotine or nicotine-containing products (eg, nicotine patch and electronic cigarette) within 3 months of screening
* Received any nonlive vaccine starting from 14 days prior to study intervention or is scheduled to receive any nonlive vaccine through 30 days following study intervention with the exception of Corona virus disease (COVID-19) vaccine administration. Study intervention must be given at least 72 hours following or at least 48 hours prior to any COVID-19 vaccination
* Consumes greater than 3 servings of alcoholic beverages per day
* Consumes excessive amounts, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, energy drinks, or other caffeinated beverages per day
* Regular user of cannabis, any illicit drugs or has a history of drug (including alcohol) abuse within approximately 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- United States (2):
  - Velocity Clinical Research, Hallandale Beach ( Site 0002), Hallandale, Florida
  - Alliance for Multispecialty Research, LLC ( Site 0001), Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 24 participants screened for inclusion, 18 participants were allocated to receive MK-0616 single dose 10-mg. All participants received at least one dose of study intervention.
Groups:
- Panel A - Moderate Renal Impairment (RI): Participants with moderate RI received a single dose of MK-616 10mg orally on Day 1.
- Panel B - Healthy Controls: Healthy matched control participants received a single dose of MK-0616 10 mg orally on Day 1.
Period: Overall Study
Arm/Group | Panel A - Moderate Renal Impairment (RI) | Panel B - Healthy Controls
Started | 10 | 8
Completed | 10 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All allocated participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Panel A - Moderate Renal Impairment (RI) | Panel B - Healthy Controls | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.5 (5.6) | 60.4 (5.0) | 63.8 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 9 | 4 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 10 | 4 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-Time Curve From Time 0 to Infinity (AUC0-Inf) of MK-0616
Description: Blood samples were collected at pre-specified timepoints to determine the AUC0-inf of MK-0616. AUC0-inf was defined as the area under the concentration-time curve of MK-0616 from time zero to infinity.
Time Frame: Predose and 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48, 72, 120, 168, 240, and 336 hours postdose
Population: All allocated participants who received a dose of study intervention and had data available for AUC0-inf.
Measure: Geometric Mean (95% Confidence Interval); unit: hour*nmol/Liter
Arm/Group | Panel A - Moderate Renal Impairment (RI) | Panel B - Healthy Controls
Number analyzed (Participants) | 7 | 6
hour*nmol/Liter | 453 [211 to 972] | 369 [211 to 646]
Statistical Analysis 1: Comparison: Panel A - Moderate Renal Impairment (RI) vs Panel B - Healthy Controls; Test type: Other — GMR: Panel A-Moderate RI/Panel B-Healthy controls; Geometric Mean Ratio (GMR) = 1.23, 90% CI 2-sided [0.62 to 2.44] — GMR and 90% confidence interval (CI) were estimated using a linear mixed effects model and referencing a t-distribution

2. Primary Outcome: Area Under the Concentration- Time Curve From Time 0 to Last Measurable Concentration (AUC0-last) of MK-0616.
Description: Blood samples were collected at pre-specified timepoints to determine the AUC0-last of MK-0616. AUC0-last was defined as the area under the concentration-time curve of MK-0616 from time zero to last measurable concentration.
Time Frame: Predose and 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48, 72, 120, 168, 240, and 336 hours postdose
Population: All allocated participants who received a dose of study intervention and had data available for AUC0-last.
Measure: Geometric Mean (95% Confidence Interval); unit: hour*nmol/Liter
Arm/Group | Panel A - Moderate Renal Impairment (RI) | Panel B - Healthy Controls
Number analyzed (Participants) | 8 | 8
hour*nmol/Liter | 312 [120 to 815] | 192 [64.1 to 574]
Statistical Analysis 1: Comparison: Panel A - Moderate Renal Impairment (RI) vs Panel B - Healthy Controls; Test type: Other — GMR: Panel A-Moderate RI/Panel B-Healthy controls; GMR = 1.63, 90% CI 2-sided [0.55 to 4.83] — GMR and 90% CI were estimated using a linear mixed effects model and referencing a t-distribution

3. Primary Outcome: Maximum Plasma Concentration (Cmax) of MK-0616
Description: Blood samples were collected at pre-specified time points to determine the Cmax of MK-0616. Cmax was defined as the maximum concentration of MK-0616 reached.
Time Frame: Predose and 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48, 72, 120, 168, 240, and 336 hours postdose
Population: All allocated participants who received a dose of study intervention and had data available for Cmax.
Measure: Geometric Mean (95% Confidence Interval); unit: nmol/Liter
Arm/Group | Panel A - Moderate Renal Impairment (RI) | Panel B - Healthy Controls
Number analyzed (Participants) | 8 | 8
nmol/Liter | 5.80 [2.98 to 11.3] | 4.00 [1.97 to 8.13]
Statistical Analysis 1: Comparison: Panel A - Moderate Renal Impairment (RI) vs Panel B - Healthy Controls; Test type: Other — GMR: Panel A-Moderate RI/Panel B-Healthy controls; GMR = 1.45, 90% CI 2-sided [0.70 to 2.99] — GMR and 90% CI were estimated using a linear mixed effects model and referencing a t-distribution

4. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) of MK-0616
Description: Blood samples were collected at pre-specified timepoints to determine the Tmax of MK-0616. Tmax was defined as time to the maximum concentration of MK-0616 reached.
Time Frame: Predose and 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48, 72, 120, 168, 240, and 336 hours postdose
Population: All allocated participants who received a dose of study intervention and had data available for Tmax.
Measure: Median (Full Range); unit: Hour
Arm/Group | Panel A - Moderate Renal Impairment (RI) | Panel B - Healthy Controls
Number analyzed (Participants) | 8 | 8
Hour | 2.00 [1.00 to 24.00] | 4.66 [1.50 to 24.02]

5. Primary Outcome: Apparent Terminal Half-life (t1/2) of MK-0616
Description: Blood samples were collected at pre-specified timepoints to determine the t1/2 of MK-0616. t1/2 was defined as the time required to divide the MK-0616 plasma concentration by two after reaching pseudo-equilibrium, following a single dose of MK-0616.
Time Frame: Predose and 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48, 72, 120, 168, 240, and 336 hours postdose
Population: All allocated participants who received a dose of study intervention and had data available for t1/2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Panel A - Moderate Renal Impairment (RI) | Panel B - Healthy Controls
Number analyzed (Participants) | 7 | 6
Hour | 55.1 (44.1) | 48.8 (32.0)

6. Primary Outcome: Apparent Clearance (CL/F) of MK-0616
Description: Blood samples were collected at pre-specified timepoints to determine the CL/F of MK-0616. CL/F was the apparent total clearance of MK-0616 in plasma over time, assessed as the rate at which MK-0616 was removed from the plasma.
Time Frame: Predose and 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48, 72, 120, 168, 240, and 336 hours postdose
Population: All allocated participants who received a dose of study intervention and had data available for CL/F.
Measure: Geometric Mean (95% Confidence Interval); unit: Liter/hour
Arm/Group | Panel A - Moderate Renal Impairment (RI) | Panel B - Healthy Controls
Number analyzed (Participants) | 7 | 6
Liter/hour | 14.2 [6.63 to 30.6] | 17.5 [9.99 to 30.5]
Statistical Analysis 1: Comparison: Panel A - Moderate Renal Impairment (RI) vs Panel B - Healthy Controls; Test type: Other — GMR: Panel A-Moderate RI/Panel B-Healthy controls; GMR = 0.82, 90% CI 2-sided [0.41 to 1.62] — GMR and 90% CI were estimated using a linear mixed effects model and referencing a t-distribution

7. Primary Outcome: Apparent Volume of Distribution (Vz/F) of MK-0616
Description: Blood samples were collected at pre-specified timepoints to determine the Vz/F of MK-0616. Vz/F was the apparent volume of distribution of MK-0616 between the plasma and the rest of the body, after dose, assessed as the total volume of MK-0616 that would need to be uniformly distributed to achieve the desired plasma drug concentration.
Time Frame: Predose and 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48, 72, 120, 168, 240, and 336 hours postdose
Population: All allocated participants who received a dose of study intervention and had data available for Vz/F.
Measure: Geometric Mean (95% Confidence Interval); unit: Liter
Arm/Group | Panel A - Moderate Renal Impairment (RI) | Panel B - Healthy Controls
Number analyzed (Participants) | 7 | 6
Liter | 1130 [675 to 1900] | 1230 [972 to 1550]
Statistical Analysis 1: Comparison: Panel A - Moderate Renal Impairment (RI) vs Panel B - Healthy Controls; Test type: Other — GMR: Panel A-Moderate RI/Panel B-Healthy controls; GMR = 0.92, 90% CI 2-sided [0.60 to 1.42] — GMR and 90% CI were estimated using a linear mixed effects model and referencing a t-distribution

8. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. Number of participants who experienced an AE were reported.
Time Frame: Up to approximately 14 days
Population: All allocated participants who received a dose of intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Panel A - Moderate Renal Impairment (RI) | Panel B - Healthy Controls
Number analyzed (Participants) | 10 | 8
Participants | 3 | 2

9. Secondary Outcome: Number of Participants Who Discontinued From the Study Due to an AE
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. Number of participants who discontinued from the study due to an AE were reported.
Time Frame: Up to approximately 14 days
Population: All allocated participants who received a dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Panel A - Moderate Renal Impairment (RI) | Panel B - Healthy Controls
Number analyzed (Participants) | 10 | 8
Participants | 0 | 0

10. Secondary Outcome: Amount Recovered in Urine From 0 to 24 Hours (Ae0-24) of MK-0616
Description: Urine samples were collected at pre-specified time points to determine the AE0-24 of MK-0616. Ae0-24 was defined as the amount of MK-0616 recovered in urine from time 0-24 hours.
Time Frame: Predose and at 0, 4, 8, 12 and 24 hours postdose
Population: All allocated participants who received a dose of study intervention and had data available for Ae0-24.
Measure: Geometric Mean (95% Confidence Interval); unit: Miligram
Arm/Group | Panel A - Moderate Renal Impairment (RI) | Panel B - Healthy Controls
Number analyzed (Participants) | 10 | 7
Miligram | 0.0116 [0.00288 to 0.0467] | 0.0141 [0.00485 to 0.0409]
Statistical Analysis 1: Comparison: Panel A - Moderate Renal Impairment (RI) vs Panel B - Healthy Controls; Test type: Other — GMR: Panel A-Moderate RI/Panel B-Healthy controls; GMR = 0.82, 90% CI 2-sided [0.22 to 3.10] — GMR and 90% CI were estimated using a linear mixed effects model and referencing a t-distribution

11. Secondary Outcome: Fraction of Dose Recovered in Urine (Fe) of MK-0616
Description: Urine samples were collected at pre-specified time points to determine the Fe of MK-0616. Fe was defined as the fraction of dose of MK-0616 recovered in urine.
Time Frame: Predose and at 0, 4, 8, 12, 24, 36 and 48 hours postdose
Population: All allocated participants who received a dose of study intervention and had data available for Fe.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent
Arm/Group | Panel A - Moderate Renal Impairment (RI) | Panel B - Healthy Controls
Number analyzed (Participants) | 10 | 7
Percent | 0.116 [0.0288 to 0.467] | 0.141 [0.0485 to 0.409]
Statistical Analysis 1: Comparison: Panel A - Moderate Renal Impairment (RI) vs Panel B - Healthy Controls; Test type: Other — GMR: Panel A-Moderate RI/Panel B-Healthy controls; GMR = 0.82, 90% CI 2-sided [0.22 to 3.10] — GMR and 90% CI were estimated using a linear mixed effects model and referencing a t-distribution

12. Secondary Outcome: Renal Clearance (CLr) of MK-0616
Description: Urine samples were collected at pre-specified time points to determine the CLr of MK-0616. was defined as the time it takes for the MK-0616 to be completely removed by the kidneys.
Time Frame: Predose and 4, 8, 12, 24, 36, and 48 hours postdose
Population: All allocated participants who received a dose of study intervention and had data available for CLr.
Measure: Geometric Mean (95% Confidence Interval); unit: Liter/hour
Arm/Group | Panel A - Moderate Renal Impairment (RI) | Panel B - Healthy Controls
Number analyzed (Participants) | 8 | 7
Liter/hour | 0.0573 [0.0157 to 0.209] | 0.152 [0.0781 to 0.294]
Statistical Analysis 1: Comparison: Panel A - Moderate Renal Impairment (RI) vs Panel B - Healthy Controls; Test type: Other — GMR: Panel A-Moderate RI/Panel B-Healthy controls; GMR = 0.38, 90% CI 2-sided [0.13 to 1.13] — GMR and 90% CI were estimated using a linear mixed effects model and referencing a t-distribution

13. Secondary Outcome: Percent Change From Baseline in Free Proprotein Convertase Subtilisin Kexin 9 (PCSK9)
Description: Urine samples were collected at pre-specified time points (baseline and 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48 and 336 hours postdose) to evaluate the reduction in free PCSK9 from baseline to up to 336 hours postdose after administration of MK-0616. The percent change from baseline in free PCSK9 was reported.
Time Frame: Baseline (Predose) and up to 336 hours post dose
Population: All allocated participants who received a dose of study intervention, and had a baseline measure and at least one postbaseline measure of PCSK9.
Measure: Geometric Mean (90% Confidence Interval); unit: Percent Change
Arm/Group | Panel A - Moderate Renal Impairment (RI) | Panel B - Healthy Controls
Number analyzed (Participants) | 10 | 8
Percent Change
  Change from baseline to 1 hour postdose | -80.5 [-83.6 to -36.3] | -66.6 [-73.4 to -10.2]
  Change from baseline to 1.5 hours postdose | -90.9 [-97.7 to -66.2] | -88.6 [-98.3 to -54.5]
  Change from baseline to 2 hours postdose | -90.8 [-96.5 to -68.9] | -87.1 [-96.8 to -54.9]
  Change from baseline to 3 hours postdose | -89.7 [-96.1 to -67.1] | -86.0 [-95.0 to -60.7]
  Change from baseline to 5 hours postdose | -89.6 [-94.8 to -73.5] | -83.6 [-97.0 to -51.6]
  Change from baseline to 8 hours postdose | -84.9 [-91.6 to -64.3] | -78.5 [-97.8 to -35.1]
  Change from baseline to 12 hours postdose: number analyzed (Participants) | 9 | 7
  Change from baseline to 12 hours postdose | -71.8 [-80.4 to -43.5] | -60.8 [-93.4 to 9.55]
  Change from baseline to 24 hours postdose: number analyzed (Participants) | 10 | 7
  Change from baseline to 24 hours postdose | -67.2 [-75.2 to -43.8] | -27.9 [-47.3 to 6.46]
  Change from baseline to 36 hours postdose | -54.9 [-64.6 to -30.9] | 1.38 [-26.4 to 47.2]
  Change from baseline to 48 hours postdose | -44.9 [-56.6 to -15.3] | 5.11 [-10.2 to 26.2]
  Change from baseline to 336 hours postdose: number analyzed (Participants) | 10 | 5
  Change from baseline to 336 hours postdose | 5.00 [-9.22 to 27.2] | 7.50 [-4.78 to 21.2]

ADVERSE EVENTS:
Time Frame: Up to approximately 16 days
Description: All cause-mortality was reported on all allocated participants. Serious and non-serious AEs were reported for all allocated participants who received a dose of study treatment.
Groups:
- Panel A - Moderate RI: Participants with moderate renal impairment (RI) received a single dose of MK-616 10mg orally on Day 1.
Arm/Group | Panel A - Moderate RI | Panel A - Moderate Renal Impairment (RI)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 3/10 | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panel A - Moderate RI (N=10) | Panel A - Moderate Renal Impairment (RI) (N=8)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Axillary pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding thist rial 45 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/90/NCT05070390/Prot_SAP_000.pdf